CLINICAL TRIAL: NCT04376164
Title: Outcome of Low-level Laser Therapy Regarding Orthodontic Leveling and Alignment of Mandibular Anterior Segment: A Controlled Clinical Appraisal
Brief Title: Laser in Orthodontic Leveling and Alignment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tharwat osman Mohi Eldeen Elshehawy (Other)
Responsible Party: Sponsor-Investigator, Tharwat osman Mohi Eldeen Elshehawy, Dentist, Ministry of Health, MSc student, Department of Orthodontics, Faculty of Dental Medicine (Boys), Al-Azhar University, Cairo, Egypt., Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101
Record Dates: First submitted 2020-05-02; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Dental Malocclusion
Keywords: Low-level laser therapy; Orthodontic Tooth Movement; Leveling and Alignment; Little Irregularity Index.
MeSH Terms: conditions — Malocclusion | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: control group laser group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): was treated without laser intervention
- laser group (Experimental): received low level laser therapy
  Interventions: Radiation: low level laser therapy

INTERVENTIONS:
Radiation: low level laser therapy — mandibular anterior teeth were irradiated by gallium aluminum arsenide semiconductor laser with 635 nm wavelength, 6.5J/cm2energy density, for 10 seconds at 10 points (0.2 J/point) on facial and lingual aspects. This protocol was started immediately after first wire insertion and then at days 3,7,14 of the first month and repeated for additional 2 months
  Other Names: photobiomodulation
  Arms: laser group

SUMMARY:
to evaluate the outcome of LLLT regarding leveling and alignment of the mandibular anterior segment.

DETAILED DESCRIPTION:
Thirty patients, 18 females and 12 males, were included who had Class I malocclusion with moderate mandibular crowding and an average age was 19.23 ± 3.1years.They were randomly divided into two parallel groups; a control group without laser intervention and a laser group which received LLLT. All patients followed a non-extraction approach using one category of fixed appliance and matching conventional NiTi archwire sequence during 3 months observation period. In laser group, mandibular anterior teeth were irradiated by gallium aluminum arsenide semiconductor laser with 635 nm wavelength, 6.5J/cm2energy density, for 10 seconds at 10 points (0.2 J/point) on facial and lingual aspects. This protocol was started immediately after first wire insertion and then at days 3,7,14 of the first month and repeated for additional 2 months. In both groups, relief of mandibular crowding was assessed by Little's irregularity index (LII) after 4 weeks (T1), after 8 weeks (T2), and after 12 weeks (T3) intervals. Changes in LII scores were evaluated through scanned 3D models via software. In addition, the monthly rate of OTM was calculated and compared. The level of significance was set at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Selection of participants was based on the following criteria:

  1. The age range was from 15 to 25 years.
  2. All permanent teeth erupted (3rd molar not included).
  3. Angle class I occlusion with normal facial proportions.
  4. Moderate crowding in the lower dental arch assessed by Little's irregularity index that requires treatment with fixed appliance using non-extraction approach.
  5. Good oral and general health.
  6. No previous or current periodontal disease.
  7. No systemic disease or regular medication that could interfere and\or affects orthodontic teeth movement.
  8. No evidence of craniofacial anomalies, such as cleft lip and palate or previous history of trauma, bruxism or parafunction.
  9. No previous orthodontic treatment.

Exclusion Criteria:

* The patients were excluded from the study if they have:

  1. Severe crowding that requires an extraction approach.
  2. Blocked-out teeth that didn't allow for placement of the bracket at the initial bonding appointment.
  3. Poor oral hygiene or periodontally compromised teeth.
  4. Relevant medical history that interferes with orthodontic treatment.
  5. Craniofacial anomalies or previous history of trauma, bruxism or parafunction.
  6. Previous orthodontic treatment.
  7. The deep bite which interferes with orthodontic brackets placement.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the alignment rate of the mandibular anterior segment with and without low level laser therapy | 6 Months
  Effect of the LLLT on alignment of the mandibular anterior teeth through evaluation of changes in Little's Irregularity Index (LII) scores (mm) throughout 12 weeks observation period of the study

CONTACTS AND LOCATIONS:
Overall Officials: tharwat O elshehay, MSc student, Principal Investigator — Al-Azhar University
Locations (1):
- Al-Azhar university, Cairo, Egypt